CLINICAL TRIAL: NCT02513875
Title: Prevention of Type 2 Diabetes in Women With Prediabetes Using Vitamin D Supplementation and Lifestyle Intervention in North India (PREVENT-WIN Study)
Brief Title: Prevention of Type 2 Diabetes With Vitamin D
Acronym: PREVENT-WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Principal Investigator, Dr Anoop Misra, Principal Investigator, Diabetes Foundation, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PREVENT-WIN 2012
Record Dates: First submitted 2015-07-29; First posted 2015-08-03 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2012-07

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D with diet and lifestyle (Experimental): vitamin D supplementation along with diet and lifestyle modification was given
  Interventions: Dietary Supplement: vitamin D
- placebo with diet and lifestyle modification (Placebo Comparator): placebo with diet and lifestyle modification was given
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D — 60,000 IU per week for 8 weeks
  Arms: vitamin D with diet and lifestyle
Dietary Supplement: Placebo — placebo +diet and lifestyle
  Arms: placebo with diet and lifestyle modification

SUMMARY:
The work plan will have the following S&T components. Component 1: Cross-sectional Study

Cross-sectional study will be of 1.5 years where 400 women from rural will be screened randomly for the vitamin D deficiency and its determinants including duration of sun exposure.

Component 2: Prospective Study

This open-label randomized placebo-controlled trial would be done in 150 pre-diabetic women with vitamin D deficiency. The women will be recruited from cross-sectional study, out patient department and health camps and they will be followed up for 2 years. The women will be randomized into two groups; lifestyle modification counseling along with intervention with either vitamin D or placebo. The levels of vitamin D and blood glucose will be assessed periodically (every 6 months). In those having recurrent vitamin D deficiency, the course of vitamin D will be repeated. At the end of the study, incidence of T2DM in both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 20-60 years.

Exclusion Criteria:

* Received Vitamin D or calcium supplementation in the previous six months.
* On any medication within last one month which could potentially influence insulin secretion, insulin sensitivity, vitamin D or calcium metabolism (e.g. metformin, thiazolidenediones, steroids etc.) and on any medication that activate steroid and xenobiotic receptors, and drugs used in transplantation
* Pregnancy and lactation at time of study
* Severe end organ damage or chronic diseases: renal/hepatic failure, any malignancy, major systemic illness etc.
* Known case of HIV infection.
* Known case of diabetes mellitus and other endocrine disorders.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
fasting glucose (mg/dL) | 2 years

SECONDARY OUTCOMES:
TC (mg/dL) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, Principal Investigator — Diabetes Foundation, India
Locations (1):
- Fortis CDOC center of Excellence for Diabetes Obesity and Endocrinoogy, New Delhi, India, Delhi, India